CLINICAL TRIAL: NCT04260945
Title: CD19/CD20 Dual-CAR-T for Patients With B-cell Leukemia
Brief Title: CD19/CD20 Dual-CAR-T in B-cell Leukemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-007
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-08

CONDITIONS: B-cell Leukemia
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD20 Dual-CAR-T cells (Experimental): CD19/CD20 Dual-CAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of CAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 250mg/m2 for 3 days and take a rest for 2 days before infusion.
  Interventions: Biological: CD19/CD20 Dual-CAR-T cells

INTERVENTIONS:
Biological: CD19/CD20 Dual-CAR-T cells — CD19/CD20 Dual-CAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of CAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 250mg/m2 for 3 days and take a rest for 2 days before infusion.CD19/CD20 Dual-CAR-T cells will be intravenously infused with a escalated dose of 0.6-3×106 cells/kg.

SUMMARY:
This is a single center, single arm, open-label, phase I study to evaluate the safety and efficacy of CD19/CD20 Dual-CAR-T cells in patients with refractory and relapsed B-cell leukemia.

DETAILED DESCRIPTION:
This Phase I study is designed as a pilot trial evaluating the safety and efficacy of CD19/CD20 Dual-CAR-T cell therapy in subjects with refractory and relapsed B cell leukemia. Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of CD19/CD20 Dual-CAR-T cells. Safety and efficacy of CD19/CD20 Dual-CAR-T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19/CD20 Dual-CAR-T cells therapy in patients with refractory and relapsed B-cell leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed and refractory B-cell acute malignancies with:

   * Relapsed after competed remission, could not get competed remission after at more than 1 course of chemotherapy (including MRD≥0.1%);
   * MRD≥0.1% after allogeneic hematopoietic stem cell transplantation(HSCT), or recurrence after complete remission or MRD ≥ 0.1% after HSCT;
   * Refractory: at least two courses of chemotherapy did not achieve complete remission or MRD ≥ 0.1%;
2. Patients must have evaluable evidence of disease, including minimal residual disease (MRD);
3. Ph + patients who meet the following criteria can register:Failure to tolerate TKI or TKI treatment failure, or failure to transplant;
4. Double positive expression of CD19 / CD20 in B cells;
5. Ages 1 to 70 years, including boundary values;
6. ECOG score 0-3 points;
7. Women of childbearing age (15-49 years old) must receive a pregnancy test within 7 days prior to initiation of treatment and the results are negative; male and female patients with fertility must use an effective contraceptive to ensure 3 months after discontinuation of treatment during the study period not pregnant inside.
8. Patients who voluntarily sign informed consent and are willing to comply with treatment plans.

Exclusion Criteria:

1. patients with organ failure:

   * Heart: NYHA heart function grade IV;
   * Liver: Grade C that achieves Child-Turcotte liver function grading;
   * Kidney: kidney failure and uremia;
   * Lung: symptoms of respiratory failure;
   * Brain: a person with a disability;
2. Active infections that are difficult to control;
3. Human immunodeficiency virus (HIV) positive;
4. Liver and kidney function: total bilirubin > 5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 5 × ULN, serum creatinine clearance rate 60mL / min;
5. GVHD ≥ 2 or anti-GVHD treatment;
6. Received allogeneic cell therapy within 4 weeks, such as donor lymphocyte infusion;
7. Subject received anti-tumor treatment (chemotherapy, mAb, or hormone) for less than 1 week;
8. Central nervous system white blood that is symptomatic or uncontrolled by systemic chemotherapy and intrathecal chemotherapy (a large number of tumor cells in CSF, white blood cell count >15WBCs/mL);
9. intracranial hypertension or unconsciousness; respiratory failure; diffuse vascular internal coagulation;
10. pregnant or lactating women;
11. The patient does not agree to use effective contraception during the treatment period and for the next 3 months;
12. Patients who participate in other clinical studies at the same time;
13. The investigator believes that there are other factors that are not suitable for inclusion or influence the subject's participation or completion of the study.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events. | 6 months
Objective remission rate(ORR) | 6 months
  The percentage of participants who achieved complete remission (CR) and partial remission over all participants.

SECONDARY OUTCOMES:
Relapse-Free Survival(RFS ) | 6 months
Overall-Survival(OS) | 6 months
Persistence of CAR-T cells in vivo | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China